CLINICAL TRIAL: NCT05391971
Title: A Randomized, Double Blind, Placebo-controlled Study of the Effects of Stellate Ganglion Block on Neural Activity and Symptoms in Participants With Post-traumatic Stress Disorder
Brief Title: Effects of Stellate Ganglion Block in Post-traumatic Stress Disorder
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-00374
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stellate Ganglion Block (SGB) Group (Experimental)
  Interventions: Drug: Bupivacaine
- Control Group (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — At the C6 level, a total of 7cc of 0.5% bupivacaine will be injected slowly at this level, with negative aspiration every 2cc. The same procedure will be repeated at the C4 level directed towards the upper cervical ganglion ventral to the longus colli muscle with a total of 3cc of 0.5% bupivacaine.
  Other Names: Marcaine
  Arms: Stellate Ganglion Block (SGB) Group
Drug: Saline — At the C6 level, a total of 7cc of saline control will be injected slowly at this level, with negative aspiration every 2cc. The same procedure will be repeated at the C4 level directed towards the upper cervical ganglion ventral to the longus colli muscle with a total of 3cc of saline control.
  Arms: Control Group

SUMMARY:
This study will enroll patients meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for post-traumatic stress disorder (PTSD). Following an initial screening visit, clinical assessment, and enrollment, subjects will be randomized into treatment and placebo arms. Both cohorts will undergo a pre-intervention functional magnetic resonance imaging (fMRI) of their brain. Treatment subjects will receive unilateral two-level stellate ganglion block via ultrasound-guided injection of anesthetic (bupivacaine) into the cervical sympathetic tissue; placebo subjects will receive an identical volume of saline via the same procedures.

At approximately 4 weeks post-procedure, both cohorts will then undergo a post-intervention clinical assessment. Finally, both cohorts will undergo a post-intervention fMRI of their brain.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. Chronic (at least one month post-trauma) DSM-5 PTSD symptoms
3. CAPS-5 Past Month score ≥ 26
4. Meets current DSM-5 PTSD diagnosis
5. Stable medications for 3 or more months by the time of study entrance (with the exception of benzodiazepines)
6. Willing and able to provide informed consent

Exclusion Criteria:

1. History of stellate ganglion block treatment
2. Allergy to local anesthetics (e.g. ropivacaine, bupivacaine)
3. Allergy to iodinated contrast agents
4. Diagnosis of bipolar I disorder with a past year manic episode
5. Diagnosis of a psychotic disorder or psychotic symptoms
6. Diagnosis of current moderate or severe substance use disorder
7. History of neurological disease (that involves the brain), seizure, or significant head trauma (i.e., extended loss of consciousness, neurological sequelae, or known structural brain lesion)
8. Significant recent suicidal ideation or significant suicidal behavior in the past 12 months or suicidal ideation with imminent risk that warrants a higher level of care
9. Concurrent trauma focused psychotherapy
10. Pregnancy (to be ruled out by urine ß-HCG)
11. Metallic implants or devices contraindicating magnetic resonance imaging by interfering with patient safety or fMRI data collection; cases will be cleared by the Principal Investigator and Center for Brain Imaging
12. Morbid obesity (BMI >4 kg/m2)
13. Current use of opioids, cocaine, or benzodiazepines (as assessed by urine toxicology)
14. Self-injurious behavior that involves suicidal intent, requires medical attention, or occurs daily.
15. Cardiac conditions or any prior heart surgeries
16. Respiratory conditions such as COPD or untreated asthma
17. History of heavy metal poisoning
18. History of neck or throat surgeries
19. Vocal cord problems or paralysis
20. Untreated high blood pressure
21. Current cancer diagnosis
22. Diagnosis of Guillain-Barré syndrome
23. Diagnosis of Parkinson's Disease
24. Unable to take 7 days off of blood thinners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Conductance Response (SCR) Amount | Week 2, Week 8
  SCR will be reported as the number of sweat glads that are activated. The more emotionally aroused an individual is, the more the SCR amount is increased. SCR will be measured during three related viewing, learning, and choice tasks, quantified as the changes between the pre-intervention fMRI scan (visit 2) and the post-intervention fMRI scan (visit 5).
Change in Cerebral Blood Flow Levels | Week 2, Week 8
  Blood flow levels will be obtained from Blood Oxygen Level Dependent (BOLD) fMRI signals during three related viewing, learning, and choice tasks, quantified as the changes between the pre-intervention fMRI scan (visit 2) and the post-intervention fMRI scan (visit 5).

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist (PCL-5) Score | Week 1
  The PCL-5 is a 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual of Mental Disorders (DSM-5) symptoms of post-traumatic stress disorder (PTSD). The self-report rating scale is 0-4 for each symptom. Rating scale descriptors are the same: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items; the higher the score, the more severe the PTSD symptoms.
Posttraumatic Stress Disorder Checklist (PCL-5) Score | Week 7
  The PCL-5 is a 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual of Mental Disorders (DSM-5) symptoms of post-traumatic stress disorder (PTSD). The self-report rating scale is 0-4 for each symptom. Rating scale descriptors are the same: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items; the higher the score, the more severe the PTSD symptoms.
Posttraumatic Stress Disorder Checklist (PCL-5) Score | Week 15
  The PCL-5 is a 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual of Mental Disorders (DSM-5) symptoms of post-traumatic stress disorder (PTSD). The self-report rating scale is 0-4 for each symptom. Rating scale descriptors are the same: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items; the higher the score, the more severe the PTSD symptoms.
Patient Health Questionnaire-9 (PHQ-9) Score | Week 1
  PHQ-9 consists of 9 items. Participants report how often they have been bothered by each item over the last 2 weeks with a score 0 (not at all) to 3 (nearly every day). The total score range is 0-27; the higher the score, the more severe the depression.
Patient Health Questionnaire-9 (PHQ-9) Score | Week 7
  PHQ-9 consists of 9 items. Participants report how often they have been bothered by each item over the last 2 weeks with a score 0 (not at all) to 3 (nearly every day). The total score range is 0-27; the higher the score, the more severe the depression.
Patient Health Questionnaire-9 (PHQ-9) Score | Week 15
  PHQ-9 consists of 9 items. Participants report how often they have been bothered by each item over the last 2 weeks with a score 0 (not at all) to 3 (nearly every day). The total score range is 0-27; the higher the score, the more severe the depression.
State-Trait Anxiety Inventory (STAI) - Form Y1 Score | Week 1
  STAI - Form Y1 is a commonly used measure of trait and state anxiety that consists of 20 statement which people have used to describe themselves. Each statement is scored from 1 (Not at all) to 4 (very much so). The total score range is 20-80; STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
State-Trait Anxiety Inventory (STAI) - Form Y1 Score | Week 7
  STAI - Form Y1 is a commonly used measure of trait and state anxiety that consists of 20 statement which people have used to describe themselves. Each statement is scored from 1 (Not at all) to 4 (very much so). The total score range is 20-80; STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
State-Trait Anxiety Inventory (STAI) - Form Y1 Score | Week 15
  STAI - Form Y1 is a commonly used measure of trait and state anxiety that consists of 20 statement which people have used to describe themselves. Each statement is scored from 1 (Not at all) to 4 (very much so). The total score range is 20-80; STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
Intolerance of Uncertainty Scale - Short Form (IUS-12) Score | Week 1
  IUS-12 is a 12-item self-report questionnaire where items are rated on 5-point Likert scales. IUS-12 is based on a definition of general uncertainty-related reactions that may be present in different anxiety disorders. Each item is scored from 1 (not at all characteristic of me) to 5 (entirely characteristic of me). The total score range is 12-60; the higher the score, the greater the intolerance of uncertainty.
Intolerance of Uncertainty Scale - Short Form (IUS-12) Score | Week 7
  IUS-12 is a 12-item self-report questionnaire where items are rated on 5-point Likert scales. IUS-12 is based on a definition of general uncertainty-related reactions that may be present in different anxiety disorders. Each item is scored from 1 (not at all characteristic of me) to 5 (entirely characteristic of me). The total score range is 12-60; the higher the score, the greater the intolerance of uncertainty.
Intolerance of Uncertainty Scale - Short Form (IUS-12) Score | Week 15
  IUS-12 is a 12-item self-report questionnaire where items are rated on 5-point Likert scales. IUS-12 is based on a definition of general uncertainty-related reactions that may be present in different anxiety disorders. Each item is scored from 1 (not at all characteristic of me) to 5 (entirely characteristic of me). The total score range is 12-60; the higher the score, the greater the intolerance of uncertainty.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Glimcher, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the data upon reasonable request. Requests should be directed to paulg@nyu.edu. To gain access, data requestors will need to sign a data access agreement.